CLINICAL TRIAL: NCT02273531
Title: Bioequivalence of a New Asasantin Capsule Formulation (Extended Release Combination 200 mg Dipyridamole/25 mg ASA) Compared to the Commercially Available Asasantin Capsule Formulation (Aggrenox®; Extended Release Combination 200 mg Dipyridamole/25 mg ASA) Following Multiple Oral Administration at Steady State After a run-in Phase (Persantine ER BID for 2 Days Each: 25 mg, 50 mg, 100 mg, 150 mg [Persantine®]; 200 mg Dipyridamole/25 mg ASA [Asasantin ER])- an Open Label, Randomized, Multiple-dose, Two-way Crossover, Change-over Study in Healthy Male and Female Volunteers
Brief Title: Bioequivalence of a New Asasantin Formulation Extended Release (ER) Compared to the Commercially Available Asasantin Formulation (Aggrenox®; Extended Release) in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9.149
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Aspirin, Dipyridamole Drug Combination

ARMS (2):
- Asasantin ER, new formulation (Experimental)
  Interventions: Drug: Asasantin ER, new formulation
- Asasantin ER, present commercial formulation (Active Comparator)
  Interventions: Drug: Asasantin ER, present commercial formulation

INTERVENTIONS:
Drug: Asasantin ER, new formulation
  Arms: Asasantin ER, new formulation
Drug: Asasantin ER, present commercial formulation
  Other Names: Aggrenox®
  Arms: Asasantin ER, present commercial formulation

SUMMARY:
Study to establish the bioequivalence of a new formulation of Asasantin ER compared to the present commercially available Asasantin ER formulation (Aggrenox®)

ELIGIBILITY:
Inclusion Criteria:

* Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead ECG, clinical laboratory tests:

  * No finding deviating from normal and of clinical relevance
  * No evidence of a clinically relevant concomitant disease
* Age ≥ 21 and ≤ 65 years
* Body mass index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and the local legislation
* Able to communicate well with the investigator and to comply with study requirements

Exclusion Criteria:

* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 14 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on trial days Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre
* History of frequent headaches
* History of gastro-intestinal ulcer disease

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. oral contraceptives, sterilization, intrauterine device (IUD)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-01; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of dipyridamole in plasma over one dosing interval at steady state (AUCτ,ss) | up to 17 days
Maximum measured concentration of dipyridamole in plasma at steady state (Cmax,ss) | up to 17 days

SECONDARY OUTCOMES:
Minimum measured concentration of dipyridamole in plasma at steady state (Cmin,ss) | up to 17 days
Average concentration of dipyridamole in plasma at steady state (Cavg) | up to 17 days
Time from dosing to the maximum concentration of dipyridamole in plasma at steady state (tmax,ss) | up to 17 days
Peak trough fluctuation of dipyridamole in plasma (PTF) | up to 17 days
Amount of the analytes that were eliminated in urine (Ae) | up to 24 hours after drug administration
Fraction in percent of dose of the analytes that was eliminated in urine (fe) | up to 24 hours after drug administration
Number of subjects with clinically significant changes in 12-lead ECG | up to 17 days
Number of subjects with clinically significant changes in vital signs (blood pressure, pulse rate) | up to 17 days
Number of subjects with clinically significant changes in laboratory tests | up to 17 days
Number of subjects with adverse events | up to 17 days
Assessment of tolerability by the investigator on a 4-point scale | after 17 days